CLINICAL TRIAL: NCT01615237
Title: Implementing Tobacco Use Treatment Guidelines in Dental Public Health Clinics
Brief Title: Dentistry United to Extinguish Tobacco
Acronym: DUET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-01148
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Tobacco Use Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBP + PF (Active Comparator): Field sites randomly assigned to Arm 2 will receive as an intervention current best practices and quarterly audits and performance feedback reports (PF) on provider delivery of cessation services using chart audit procedures that we have used successfully in prior work. Depending on what is used at the site, paper or Electronic Dental Record, we will work with the site to create a registry of patients who are tobacco users.
  Interventions: Behavioral: Audit and performance feedback (PF); Behavioral: Current Best Practices (CBP)
- CBP + PF + P4P (Active Comparator): Field sites randomly assigned to this implementation condition (Arm 3) will receive current best practices (CBP), quarterly audit and performance feedback reports (PF), and financial incentives (pay for performance, P4P) for every documented (documentation in patient chart of counseling, prescription, or referral to the quit-line) delivery of adherence to clinical practice guidelines.
  Interventions: Behavioral: Audit and performance feedback (PF); Behavioral: Financial Incentive (P4P); Behavioral: Current Best Practices (CBP)
- Current Best Practices (CBP) (Active Comparator): All dental field sites will receive current best practices (CBP) for training and technical assistance in promoting adoption of clinical practice guidelines for treating tobacco dependence.
  Interventions: Behavioral: Current Best Practices (CBP)

INTERVENTIONS:
Behavioral: Audit and performance feedback (PF) — Quarterly, trained clinic staff will use a standardized chart audit tool to evaluate documentation of cessation assistance. The feedback report will show individual and clinic performance summaries of two targeted provider behaviors based on documentation in the chart: 1) percentage of smokers advised to quit, and 2) percentage of smokers who received quitting assistance. Quitting assistance will be fulfilled by documentation of any of the following provider behaviors: a) Faxing a referral to the New York State (NYS) Quitline, b) Chart documentation of providing cessation counseling; and/or c) discussing and or prescribing cessation medications. Reports will be given to the Dental Director, who will be instructed to distribute them to dental providers no later than 30 days following the end of the quarter.
  Arms: CBP + PF; CBP + PF + P4P
Behavioral: Financial Incentive (P4P) — We will review charts of all smokers to evaluate documentation of cessation assistance (i.e., prescription given for cessation medication, the provision of brief cessation counseling and/or a fax referral to the NYS Quitline or other local cessation support program). Sites will receive $20 for each patient with chart documentation of receiving tobacco cessation assistance. The P4P reimbursement will be offered quarterly with an annual cap of $5000 to each site as employees are salaried.
  Arms: CBP + PF + P4P
Behavioral: Current Best Practices (CBP) — CBPs that will be implemented is consistent with the PHS recommended guidelines and is as follows: The dental care team will assess smoking status, deliver advice to quit, assess readiness to quit, provide patient education materials, a prescription for cessation pharmacotherapy and referral to the NYS Quitline, and document findings and treatment plan on the chart system. In New York State, the Quitline provides free medication for uninsured. As brief provider interventions have been shown to be effective, the recommended tobacco treatment protocol will require approximately 5-10 minutes.

SUMMARY:
System level strategies for implementing tobacco use treatment guidelines exist but are insufficiently put into practice, particularly in dental care settings. Closing the gap between research and practice is stymied by the limited research on systems changes necessary to implement tobacco treatment in routine dental care. Drawing from a burgeoning dissemination science literature, the proposed study compares the cumulative benefit of the following three systems-level strategies: 1) staff training and clinical reminders, 2) provider feedback and 3) pay-for- performance (financial incentives), that have been widely endorsed by a 2001 Institute of Medicine Report, "Crossing the Quality Chasm" (IOM 2011) and the 2008 PHS Guidelines (Fiore 2007, Fiore 2008, IOM 2011).

The investigators propose a 3-arm cluster randomized controlled trial that will analyze the implementation process and compare the cost and effectiveness of three implementation strategies: 1) Staff training and CBP in implementing PHS Guidelines; 2) CBP + provider performance feedback (PF) and 3) CBP + PF + Pay-for-performance (provider reimbursement for tobacco cessation treatment delivery). Guided by Organizational Change Theory and the Theory of Planned Behavior (Ajzen 1991, Damschroder 2009, Greenhalgh 2004, Solberg 2007) the investigators will identify multi-level factors that facilitate or impede the implementation process in dental clinics. Our primary outcome is improvement in provider delivery of tobacco cessation treatment found through extensive meta-analysis (Fiore 2008) to be an essential determinant of patient cessation outcomes. Our secondary outcome will be post-intervention patient-reported quit rates. In addition to examining the comparative effectiveness of the three implementation strategies, the investigators will use a mixed methods approach to examine implementation processes (Aim 2) to assess the degree to which the interventions are integrated into practice as intended and to clarify the mechanisms through which the intervention influences provider behavior.

DETAILED DESCRIPTION:
Purpose of the Study System level strategies for implementing tobacco use treatment guidelines exist but are insufficiently put into practice, particularly in dental care settings. Closing the gap between research and practice is stymied by the limited research on systems changes necessary to implement tobacco treatment in routine dental care. Drawing from a burgeoning dissemination science literature, the proposed study compares the cumulative benefit of the following three systems-level strategies: 1) staff training and clinical reminders, 2) provider feedback and 3) pay-for- performance (financial incentives), that have been widely endorsed by a 2001 Institute of Medicine Report, "Crossing the Quality Chasm" (IOM 2011) and the 2008 PHS Guidelines (Fiore 2007, Fiore 2008, IOM 2011).

Staff Training and Clinical Reminder Systems. The PHS Guideline strongly recommends staff training, clinical reminder systems and other practice supports as the foundation for treating tobacco dependence in health care settings. Despite observed limitations (Curry 2008, Grimshaw 2003, Shelley 2010), staff training, practice supports, clinical reminder systems and referral pathways represent current best practices (CBP) for screening and treating tobacco dependence.

Performance Feedback (PF). In recent randomized trials conducted in primary medical care settings, clinical audit and feedback with regard to tobacco treatment performance have been associated with a twofold increase in cessation assistance and referral to cessation quitlines (Bentz 2007, Curry 2008, Wadland 2007). While clinical audit and feedback have been shown to increase provider adherence to tobacco use treatment guidelines in medical settings, these strategies have not yet been examined in dental practice (Curry 2000, Curry 2008, Fiore 2007, Fiore 2008, Grimshaw 2006, Solberg 2000).

Pay for Performance (P4P). P4P or providing financial incentives for meeting predetermined performance goals has attracted much interest as a strategy to improving guideline implementation and the quality of care (Petersen 2006, Sonnad, 1998). The recent consensus report from the 2nd European Workshop on Tobacco use Prevention and Cessation for Oral Health Professionals emphasized the importance of appropriate compensation of tobacco use treatment to provide incentive to oral health providers (Ramseier 2010). Several studies have demonstrated a positive association between P4P and adherence to recommended tobacco use treatment (An 2008, Coleman, 2010, Roski, 2003). For instance, An et al, found that a P4P program increased referrals to statewide tobacco quitline services (An 2008). Electronic dental records and automated billing systems (such as the Dentrix system used by most of our participating dental clinic sites) are adding nicotine dependence diagnostic and treatment procedure codes. This health informatics trend bodes well for the sustainability of performance feedback and P4P implementation strategies.

Background Based on meta-analyses of over 8000 tobacco cessation studies published in the past three decades, the 2008 Public Health Service (PHS) Guideline, Treating Tobacco Use and Dependence provides strong evidence that provider delivery of tobacco dependence treatment, including cessation pharmacotherapy and brief counseling, can produce significant and sustained reductions in tobacco use and should be delivered to all smokers seeking routine health care (Fiore 2008). Provider adherence to the PHS Guideline recommendations requires Asking all patients about tobacco use, Advising smokers to quit, Assessing readiness to quit, providing cessation Assistance and Arranging follow-up (5As) (Fiore 2008). Adequate implementation of the PHS Guidelines would generate 1.6 million additional quitters per year and nearly 3.3 million quality life years saved (USDHHS 2000).

Despite the existence of effective tobacco dependence treatments, inadequate adoption, particularly among low income and ethnic/racial minority smokers, has contributed to growing disparities in smoking prevalence and tobacco-related illness (Fagan, 2007, King 2010, Lopez-Quintero 2006). For instance, Hispanics are 57% and African-Americans 13% less likely to receive physician advice to quit than non-Hispanic whites (Lopez-Quintero 2006). Citing persistent missed opportunities to promote tobacco cessation, the Institute of Medicine's (IOM) report, "Ending the Tobacco Problem: A Blueprint for the Nation", calls for greater efforts to implement effective tobacco cessation interventions in health care settings. The USDHHS Task Force on Tobacco Control recently highlighted the need to better understand provider incentives and other system-level strategies to motivate provider adherence to PHS guidelines and leverage emerging opportunities for reimbursement of preventive services as presented by the 2010 Affordable Care Act. These recent health policy reports highlight the need and potential public health value of reducing tobacco-related disparities through dissemination of evidence-based interventions in health care delivery systems serving low income and other high-risk smokers (Medicine. lo 2007, Services US Department of Health and Human Services 2010).

Dental care settings have several advantageous features for delivery of tobacco cessation treatment including: 1) broad reach with 62.8% of 18-64 years olds reporting at least one annual dental visit (Manski 2007), 2) access to patients who do not receive other healthcare services (10% of dental patients do not regularly see a physician) (Strauss 2006), 3) the dental team routinely provides preventive services; and 4) controlled trials have demonstrated the efficacy of dental office-based cessation interventions (Gordon 2006). Moreover, dental professionals have a credible role in providing tobacco cessation treatment in view of the oral hazards of tobacco use. A recent national survey found that 88.7% of dentists and 96% of dental hygienists reported that treating tobacco use was an important professional responsibility (Tong 2010). Although most dentists still work in private practice settings, there are about 475 federally-funded, community or neighborhood health centers with dental clinics and another 250 community dental clinics throughout the United States (Gordon 2005). These community dental health centers serve predominantly low income populations known to have a high prevalence of smoking (Gordon 2010). Therefore, the potential impact of implementing the Tobacco Guidelines in these public health dental clinics is substantial (Gordon 2006). Unfortunately, delivery of tobacco use treatment in routine dental care remains limited (Albert 2002, Albert 2005, Tong 2010).

Although national surveys indicate that dental providers are increasingly screening for tobacco use and offering brief advice, adherence to the PHS guidelines in inconsistent with only 10-25% dental health professionals' routinely delivering cessation assistance (e.g. cessation pharmacotherapy prescriptions and/or referral for cessation counseling) (Albert 2002, Tong 2010). Dentists most often cite lack of training, and adequate reimbursement to explain their subpar performance in providing tobacco cessation interventions (Albert 2005). Challenges to wide-scale implementation of tobacco dependence treatment also include a lack of referral resources and a lack of office-based systems (Gordon 2006, Albert 2005). PHS guideline implementation is likely affected by both provider attitudes and organizational priorities that impact provider behavior (Albert 2002, Curry 2000, Fiore 2008).

Study Design We propose a 3-arm cluster randomized controlled trial that will analyze the implementation process and compare the cost and effectiveness of three implementation strategies: 1) Staff training and CBP in implementing PHS Guidelines; 2) CBP + provider performance feedback (PF) and 3) CBP + PF + Pay-for-performance (provider reimbursement for tobacco cessation treatment delivery). Guided by Organizational Change Theory and the Theory of Planned Behavior (Ajzen 1991, Damschroder 2009, Greenhalgh 2004, Solberg 2007) we will identify multi-level factors that facilitate or impede the implementation process in dental clinics. Our primary outcome is improvement in provider delivery of tobacco cessation treatment found through extensive meta-analysis (Fiore 2008) to be an essential determinant of patient cessation outcomes. Our secondary outcome will be post-intervention patient-reported quit rates. In addition to examining the comparative effectiveness of the three implementation strategies, we will use a mixed methods approach to examine implementation processes (Aim 2) to assess the degree to which the interventions are integrated into practice as intended and to clarify the mechanisms through which the intervention influences provider behavior.

Clinic level selection of performance sites is guided by our desire to ensure that our findings would be generalizable to real-world dental health care settings serving diverse population of smokers. We will partner with 18 public health dental clinics that have expressed willingness to participate. For practical (cost and staffing) reasons, we will recruit clinics in six successive waves with three sites enrolled per wave (see Timeline). Clinic randomization will be conducted by the Memorial Sloan Kettering Cancer Center Clinical Research Database Program (CRDB) within the Biostatistics Service using the random permuted block method.

ELIGIBILITY:
Inclusion Criteria:

* Clinics are included if they are located within the NYC metropolitan area and employ at least three FTE dentists.
* Providers are included if they practice full-time or part-time at one of the study clinics
* Patients are included if they are 18 years or older, active smokers defined as those who report smoking cigarettes some days, most days, or every day and have smoked in the past 7 days, have an appointment with a dentist or hygienist, NYS resident, speak English, Spanish, Chinese or Russian, and are able to comply with study procedures in the opinion of the principal investigator.

Exclusion Criteria:

* Clinic locations are excluded if the number of unique adult patient visits per week averages less than 100, if the dental director reports that the clinic assists more than 60% of patients with tobacco cessation and if the clinics policies would prohibit the clinic from accepting pay-for-performance funds if randomized to that arm. All sites with less than 3 dental providers will also be excluded.
* Providers are excluded if they do not speak English.
* Patients are excluded if they do not speak English, Spanish, Chinese or Russian, and if they have already completed the patient exit interview during the same intervention phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3207 (Actual)
Dates: Start 2013-03-09 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
To assess the primary outcome of provider adherence to tobacco use treatment guidelines, we will conduct patient exit interviews with 80 smokers pre and post-intervention at each of the 18 study sites (2880 smokers pre and post). | prior to and approximately 12 months following each site's enrollment in the study
  The Patient Exit Interview (PEI) is a brief patient-reported measurement tool for the assessment of provider delivery of tobacco use treatment. Patients will be approached during their clinic visits by trained research study assistants, to determine smoking status and to obtain consent. Patient eligibility includes: 1) age 18 or over; and 2) active smokers defined as those who report smoking within the past 7 days.
Compare the effectiveness of the three intervention arms on provider behavior for aiding patient's tobacco cessation | June 2013-June 2017
  We will also conduct provider surveys with all participating dentists and dental directors, and focus groups with all participating dental providers, dental directors and other key informants, including stakeholders in administrative and technical roles before and after the intervention.
  For the provider surveys, we will be asking all the dental providers (dental directors, dentists, dental hygienists, dental residents) to complete the surveys. We expect to enroll approximately 30 providers at each site for a total of 540 providers for the provider surveys. The number of participating dentists from each site will vary depending upon the size of the dental practice.

SECONDARY OUTCOMES:
Cost analysis | last two years of the study/ end of each site's enrollment period
  We will separate estimate research costs (e.g. labor and other inputs associated with grant administration, Institutional Review Board approval, manuscript prep) and direct clinical intervention costs (e.g. dental provider time associated with counseling patients, staff training, IT costs, reimbursement costs). The New York State Quitline has estimates of their counseling cost per quit.
assess patient utilization of cessation services and smoking abstinence | 0-6 months post intervention phase
  We will capture patient reported quit rates and utilization of cessation services on the post-intervention Patient Exit Interview

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, MD, MPH, Principal Investigator — NYU Langone Health; Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Background] Albert DA, Severson H, Gordon J, Ward A, Andrews J, Sadowsky D. Tobacco attitudes, practices, and behaviors: a survey of dentists participating in managed care. Nicotine Tob Res. 2005 Apr;7 Suppl 1:S9-18. doi: 10.1080/14622200500078014. PMID 16036273
- [Background] Albert D, Ward A, Ahluwalia K, Sadowsky D. Addressing tobacco in managed care: a survey of dentists' knowledge, attitudes, and behaviors. Am J Public Health. 2002 Jun;92(6):997-1001. doi: 10.2105/ajph.92.6.997. PMID 12036795
- [Background] An LC, Bluhm JH, Foldes SS, Alesci NL, Klatt CM, Center BA, Nersesian WS, Larson ME, Ahluwalia JS, Manley MW. A randomized trial of a pay-for-performance program targeting clinician referral to a state tobacco quitline. Arch Intern Med. 2008 Oct 13;168(18):1993-9. doi: 10.1001/archinte.168.18.1993. PMID 18852400
- [Background] Bentz CJ, Bayley KB, Bonin KE, Fleming L, Hollis JF, Hunt JS, LeBlanc B, McAfee T, Payne N, Siemienczuk J. Provider feedback to improve 5A's tobacco cessation in primary care: a cluster randomized clinical trial. Nicotine Tob Res. 2007 Mar;9(3):341-9. doi: 10.1080/14622200701188828. PMID 17365766
- [Background] Coleman T. Do financial incentives for delivering health promotion counselling work? Analysis of smoking cessation activities stimulated by the quality and outcomes framework. BMC Public Health. 2010 Mar 26;10:167. doi: 10.1186/1471-2458-10-167. PMID 20346154
- [Background] Curry SJ, Keller PA, Orleans CT, Fiore MC. The role of health care systems in increased tobacco cessation. Annu Rev Public Health. 2008;29:411-28. doi: 10.1146/annurev.publhealth.29.020907.090934. PMID 18173387
- [Background] Curry SJ. Organizational interventions to encourage guideline implementation. Chest. 2000 Aug;118(2 Suppl):40S-46S. doi: 10.1378/chest.118.2_suppl.40s. PMID 10939998
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Fagan P, Moolchan ET, Lawrence D, Fernander A, Ponder PK. Identifying health disparities across the tobacco continuum. Addiction. 2007 Oct;102 Suppl 2:5-29. doi: 10.1111/j.1360-0443.2007.01952.x. PMID 17850611
- [Background] Clinical Practice Guideline Treating Tobacco Use and Dependence 2008 Update Panel, Liaisons, and Staff. A clinical practice guideline for treating tobacco use and dependence: 2008 update. A U.S. Public Health Service report. Am J Prev Med. 2008 Aug;35(2):158-76. doi: 10.1016/j.amepre.2008.04.009. PMID 18617085
- [Background] Gordon JS, Andrews JA, Albert DA, Crews KM, Payne TJ, Severson HH. Tobacco cessation via public dental clinics: results of a randomized trial. Am J Public Health. 2010 Jul;100(7):1307-12. doi: 10.2105/AJPH.2009.181214. Epub 2010 May 13. PMID 20466951
- [Background] Gordon JS, Andrews JA, Lichtenstein E, Severson HH. The impact of a brief tobacco-use cessation intervention in public health dental clinics. J Am Dent Assoc. 2005 Feb;136(2):179-86; quiz 230-1. doi: 10.14219/jada.archive.2005.0139. PMID 15782521
- [Background] Gordon JS, Lichtenstein E, Severson HH, Andrews JA. Tobacco cessation in dental settings: research findings and future directions. Drug Alcohol Rev. 2006 Jan;25(1):27-37. doi: 10.1080/09595230500459495. PMID 16492575
- [Background] Fiore MC, Keller PA, Curry SJ. Health system changes to facilitate the delivery of tobacco-dependence treatment. Am J Prev Med. 2007 Dec;33(6 Suppl):S349-56. doi: 10.1016/j.amepre.2007.09.001. PMID 18021910
- [Background] Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O. Diffusion of innovations in service organizations: systematic review and recommendations. Milbank Q. 2004;82(4):581-629. doi: 10.1111/j.0887-378X.2004.00325.x. PMID 15595944
- [Background] Grimshaw J, Eccles M, Thomas R, MacLennan G, Ramsay C, Fraser C, Vale L. Toward evidence-based quality improvement. Evidence (and its limitations) of the effectiveness of guideline dissemination and implementation strategies 1966-1998. J Gen Intern Med. 2006 Feb;21 Suppl 2(Suppl 2):S14-20. doi: 10.1111/j.1525-1497.2006.00357.x. PMID 16637955
- [Background] Institute of Medicine (US) Committee on Crossing the Quality Chasm: Adaptation to Mental Health and Addictive Disorders. Improving the Quality of Health Care for Mental and Substance-Use Conditions: Quality Chasm Series. Washington (DC): National Academies Press (US); 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK19830/ PMID 20669433
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: current cigarette smoking among adults aged >or=18 years --- United States, 2009. MMWR Morb Mortal Wkly Rep. 2010 Sep 10;59(35):1135-40. PMID 20829747
- [Background] Lopez-Quintero C, Crum RM, Neumark YD. Racial/ethnic disparities in report of physician-provided smoking cessation advice: analysis of the 2000 National Health Interview Survey. Am J Public Health. 2006 Dec;96(12):2235-9. doi: 10.2105/AJPH.2005.071035. Epub 2006 Jun 29. PMID 16809587
- [Background] Manski RJ, Cooper PF. Dental care use: does dental insurance truly make a difference in the US? Community Dent Health. 2007 Dec;24(4):205-12. PMID 18246837
- [Background] Petersen LA, Woodard LD, Urech T, Daw C, Sookanan S. Does pay-for-performance improve the quality of health care? Ann Intern Med. 2006 Aug 15;145(4):265-72. doi: 10.7326/0003-4819-145-4-200608150-00006. PMID 16908917
- [Background] Ramseier CA, Warnakulasuriya S, Needleman IG, Gallagher JE, Lahtinen A, Ainamo A, Alajbeg I, Albert D, Al-Hazmi N, Antohe ME, Beck-Mannagetta J, Benzian H, Bergstrom J, Binnie V, Bornstein M, Buchler S, Carr A, Carrassi A, Casals Peidro E, Chapple I, Compton S, Crail J, Crews K, Davis JM, Dietrich T, Enmark B, Fine J, Gallagher J, Jenner T, Forna D, Fundak A, Gyenes M, Hovius M, Jacobs A, Kinnunen T, Knevel R, Koerber A, Labella R, Lulic M, Mattheos N, McEwen A, Ohrn K, Polychronopoulou A, Preshaw P, Radley N, Rosseel J, Schoonheim-Klein M, Suvan J, Ulbricht S, Verstappen P, Walter C, Warnakulasuriya S, Wennstrom J, Wickholm S, Zoitopoulos L. Consensus Report: 2nd European Workshop on Tobacco Use Prevention and Cessation for Oral Health Professionals. Int Dent J. 2010 Feb;60(1):3-6. PMID 20361571
- [Background] Roski J, Jeddeloh R, An L, Lando H, Hannan P, Hall C, Zhu SH. The impact of financial incentives and a patient registry on preventive care quality: increasing provider adherence to evidence-based smoking cessation practice guidelines. Prev Med. 2003 Mar;36(3):291-9. doi: 10.1016/s0091-7435(02)00052-x. PMID 12634020
- [Background] Solberg LI. Improving medical practice: a conceptual framework. Ann Fam Med. 2007 May-Jun;5(3):251-6. doi: 10.1370/afm.666. PMID 17548853
- [Background] Solberg LI, Brekke ML, Fazio CJ, Fowles J, Jacobsen DN, Kottke TE, Mosser G, O'Connor PJ, Ohnsorg KA, Rolnick SJ. Lessons from experienced guideline implementers: attend to many factors and use multiple strategies. Jt Comm J Qual Improv. 2000 Apr;26(4):171-88. doi: 10.1016/s1070-3241(00)26013-6. PMID 10749003
- [Background] Sonnad SS. Organizational tactics for the successful assimilation of medical practice guidelines. Health Care Manage Rev. 1998 Summer;23(3):30-7. doi: 10.1097/00004010-199802330-00004. PMID 9702559
- [Background] Strauss SM, Alfano MC, Shelley D, Fulmer T. Identifying unaddressed systemic health conditions at dental visits: patients who visited dental practices but not general health care providers in 2008. Am J Public Health. 2012 Feb;102(2):253-5. doi: 10.2105/AJPH.2011.300420. Epub 2011 Dec 15. PMID 22390440
- [Background] Tong EK, Strouse R, Hall J, Kovac M, Schroeder SA. National survey of U.S. health professionals' smoking prevalence, cessation practices, and beliefs. Nicotine Tob Res. 2010 Jul;12(7):724-33. doi: 10.1093/ntr/ntq071. Epub 2010 May 27. PMID 20507899
- [Background] Wadland WC, Holtrop JS, Weismantel D, Pathak PK, Fadel H, Powell J. Practice-based referrals to a tobacco cessation quit line: assessing the impact of comparative feedback vs general reminders. Ann Fam Med. 2007 Mar-Apr;5(2):135-42. doi: 10.1370/afm.650. PMID 17389537
- [Result] Ajzen I. The theory of planned behaviour: reactions and reflections. Psychol Health. 2011 Sep;26(9):1113-27. doi: 10.1080/08870446.2011.613995. PMID 21929476
- [Derived] Ostroff JS, Li Y, Shelley DR. Dentists United to Extinguish Tobacco (DUET): a study protocol for a cluster randomized, controlled trial for enhancing implementation of clinical practice guidelines for treating tobacco dependence in dental care settings. Implement Sci. 2014 Feb 21;9:25. doi: 10.1186/1748-5908-9-25. PMID 24559178